CLINICAL TRIAL: NCT01401231
Title: Pilot Trial of Behavioral Activation Psychotherapy for Perinatal Depression
Brief Title: Behavioral Activation for Perinatal Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); HealthPartners Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: U19MH092201 (NIH); U19MH092201 (NIH)
Record Dates: First submitted 2011-07-22; First posted 2011-07-25 (Estimated); Last update posted 2017-10-13 (Actual); Status verified 2017-10

CONDITIONS: Depression During Pregnancy
Keywords: depression; pregnancy
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Behavioral Activation (Experimental): Behavioral activation psychotherapy
  Interventions: Behavioral: Behavioral activation psychotherapy
- Usual Care (Placebo Comparator): Continued care as usual
  Interventions: Other: Usual care

INTERVENTIONS:
Behavioral: Behavioral activation psychotherapy — Up to 10 sessions of behavioral activation psychotherapy delivered in person or by telephone.
  Arms: Behavioral Activation
Other: Usual care — Continued usual care (could include referral for medication or psychotherapy)
  Arms: Usual Care

SUMMARY:
This pilot study will examine the feasibility, acceptability, and effectiveness of a brief behavioral activation psychotherapy for women with perinatal depression.

ELIGIBILITY:
Inclusion Criteria:

- Pregnant PHQ9 Depression Score of 15 or greater Receiving prenatal care at one of the participating sites

Exclusion Criteria:

- Known diagnosis of bipolar or psychotic disorder Active substance dependence Immediate risk of self harm Immediate need for inpatient mental health treatment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 163 (Actual)
Dates: Start 2011-08; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
PHQ9 Depression Score | 3 months post-partm
  Mean PHQ9 depression score 3 months postpartum

CONTACTS AND LOCATIONS:
Locations (1):
- Group Health Cooperative, Seattle, Washington, United States

REFERENCES:
- [Derived] Dimidjian S, Goodman SH, Sherwood NE, Simon GE, Ludman E, Gallop R, Welch SS, Boggs JM, Metcalf CA, Hubley S, Powers JD, Beck A. A pragmatic randomized clinical trial of behavioral activation for depressed pregnant women. J Consult Clin Psychol. 2017 Jan;85(1):26-36. doi: 10.1037/ccp0000151. PMID 28045285